CLINICAL TRIAL: NCT03174626
Title: A Pilot Study on the Implementation of the WLS-Cancer Care Protocol
Brief Title: Williams LifeSkills - Cancer Caregiver Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00079526
Record Dates: First submitted 2017-05-31; First posted 2017-06-02 (Actual); Last update posted 2017-12-29 (Actual); Status verified 2017-05

CONDITIONS: Cancer
Keywords: caregiver; stress management
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WLSCC Intervention (Experimental): Williams LifeSkills framework on stress management and cancer care
  Interventions: Behavioral: WLSCC
- Usual Care (Other): No intervention is provided
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: WLSCC — Briefly, WLSCC contents are as follows: Psychosocial skill 1: Increase objectivity and awareness of thoughts and feelings in a distressing situation and learning the technique of a log entry; Psychosocial skill 2: Evaluate the situation to decide whether to change one's reactions or to take actions; Psychosocial skill 3: Increase the positive and the sense of meaning in your life; Psychosocial skill 4: Deflection strategies; Psychosocial skill 5: Take action when action is called for; Psychosocial skill 6: Assertion; Psychosocial skill 7: Saying "No"; Psychosocial skill 8 : Communication; Psychosocial skill 9: Become a better listener; Psychosocial skill 10: Empathy.
  Arms: WLSCC Intervention
Other: Usual Care — No training provided. After data collection period is over, participants have the option to receive the WLSCC training
  Arms: Usual Care

SUMMARY:
The purpose of the pilot is to test the feasibility of developing and implementing the Williams LifeSkills Cancer Care (WLSCC) and examining its preliminary impact on caregiver well-being and patient well-being. The study is a two-arm randomized intervention pilot (WLSCC vs. Usual Care [UC]) with data collection at baseline, immediately after training, and 2 weeks after completing the training. Study setting is at the breast and thoracic cancer clinics at the Duke Cancer Clinic. A total of 40 cancer patients (20 breast cancer patients and 20 lung cancer patients) and their caregivers (for a total N of 80) will be recruited for the pilot. The WLSCC will involve six 30-minute phone sessions and will encompass the application of 10 psychosocial skills within the context of cancer caregiving. Descriptive statistics will be used to detail recruitment/retention rate, fidelity rate, and the baseline demographic and clinical characteristics for the total sample and each group. Plots of the individual trajectories (within-person scores over time) will be used to identify the pattern(s) of change over time, and assess between-person variability in baseline values (intercepts) and trajectories (slopes). This study carries minimal risk to study participation.

DETAILED DESCRIPTION:
The pilot's specific aims are to:

1. Test the feasibility of (a) recruiting lung and breast cancer patients and their caregivers (hereafter, "dyads) at the Duke Cancer Center (DCC) outpatient clinic; (b) training interventionists to deliver the WLSCC protocol; (c) delivering the WLSCC protocol by phone.
2. Examine the immediate and two-week impact of the WLSCC on caregiver quality of life, anxiety and depression, caregiving preparedness, and social support as well as patient's well-being (Functional Assessment of Cancer Therapy.

Design and Procedures The pilot is two-arm randomized intervention pilot (WLSCC vs. Usual Care [UC]) with data collection at baseline (T1), immediately after training (T2), and 2 weeks after completing the training (T3). Caregivers will have an option to receive the WLCCC protocol, should they wish, after the data collection period. A stratified randomization will be conducted with stratifying variable being type of cancer and the block size will be 2.

The pilot setting is at the breast and thoracic cancer clinics at the DCC, Durham, NC. The WLSCC will involve approximately six 30-minute phone sessions between the caregiver and interventionist. The six calls will be delivered within three weeks of consent and will use intervention scripts for standardization of delivery.

The training will use the WLS format to assess issues and discuss strategies for cancer care including caregiver stress management. The context of discussion will be tailored by using the cancer issues endorsed by the cancer patient at baseline data collection. In delivering the interactive WLSCC training, the interventionist will preface each session by stating that the protocol is designed to enable them to cope more effectively with demanding caregiving situations and stressful life situations, to improve their relationships with others, and to increase the proportion of positive thoughts and feelings in their daily lives. The interventionist will frequently prompt the caregiver to raise questions that pertain to their situation (using cancer symptoms endorsed by cancer patient at baseline survey). At the end of each telephone session, the interventionist will request for the caregiver to complete log entries to provide an opportunity to reflect or put into action the WLSCC psychosocial skills taught in each session.

Subject Recruitment & Compensation:

The study team will review every week the list of adult patients who are scheduled for an outpatient visit at DCC Breast Cancer Clinic and Thoracic Clinic. For those who initially meet the criteria of aged 18 years and above and with primary breast or thoracic cancer diagnosed less than a year of the scheduled visit, the team will send an invite letter by mail to describe the study and invite their participation. A number will be provided that the patient or caregiver can call to decline participation. If no phone call or voice message is received on the opt-out number after 2 weeks of mailing the letter, the study staff will make plans to approach patient and family/friend during the visit to determine further eligibility for participation.

The study staff will visit the Duke Breast and Thoracic cancer clinic at least three times a week. She/he will approach patients who have not opted out of the study to determine if the family/friend accompanying the patient meets the definition of a caregiver for this study. If yes, the study staff will explain the study including the possibility that the dyad maybe assigned to either the WLSCC or UC group. If a working telephone number is assured and the dyads show interest in study participation, consent will be obtained from the dyad. After consent is obtained, baseline data (T1) for measures will be obtained. Using a laptop, the study staff will access study database and measures using the secure Duke server. He/she will ask questions in the baseline measures and responses will be directly entered to the study database. Thereafter, the study staff will assign the dyad a number that is randomly determined by a computer program. Each number from 1-40 will be assigned as either WLSCC or UC. The interventionist will call the caregiver at the scheduled first session. Before the first call ends, schedules for calls 2 to 6 will be established with the caregiver.

All follow-up data will be collected by phone. Follow-up data collection for T2 will be on the date of the last phone call for the WLSCC group and 3 weeks after consent was obtained in the UC group. T3 data will be collected two weeks after T2 data were collected in the WLSCC group and five weeks after consent in the UC group.

Data Analysis & Statistical Considerations:

Descriptive statistics will be used to detail recruitment/retention rate, fidelity rate, and the baseline demographic and clinical characteristics for the total sample and each group. For each caregiver and patient outcome measure, descriptive statistics will be calculated at baseline and at each follow-up. Plots of the individual trajectories (within-person scores over time) will be used to identify the pattern(s) of change over time, and assess between-person variability in baseline values (intercepts) and trajectories (slopes).Hierarchical mixed-effects models will be used to delineate and summarize trends and relationships in the data while nesting for dyads. This pilot study will focus on estimating effective size for WLSCC rather than statistical significance testing dues to the exploratory nature of the pilot study. When statistical testing is conducted, non-directional tests will be performed with level of significance set at 0.10.

ELIGIBILITY:
Inclusion Criteria:

* Patients are those with a confirmed medical diagnosis of breast or thoracic cancer regardless of stage and followed at DCC for management.
* The cancer diagnosis should have been made less than a year from the next scheduled appointment to the DCC.
* The caregiver is defined as unpaid individuals involved in assisting the cancer patient with activities of daily living and/or medical tasks.
* Patients and caregivers must be able to hear, read, and write in English; oriented to place, person, and time; and have an active telephone service, either cellular or landline.

Exclusion Criteria:

* Excluding patients and caregivers who are less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-05-03 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2017-08-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of recruitment of dyads for the WLSCC Intervention | 6 months
  Feasibility of recruiting as measured by the number of dyads approached per clinic visit
Feasibility of agreeing to participate in the WLSCC study | 6 months
  Feasibility of recruiting as measured by the number of yes vs no to study participation
Feasibility of participating in phone calls for the study | 6 months
  Feasibility of recruiting as measured by the rate of participation in phone calls
Feasibility of recruitment and completion of measures | 6 months
  Feasibility of recruiting as measured by the completion of outcome measures including baseline demographics (please see below under secondary outcome measures for list of outcome measures)
Feasibility of recruitment longevity for the WLSCC Intervention | 6 months
  Feasibility of recruiting as measured by the attrition rate at the end of data collection
Feasibility of recruitment for the WLSCC study for control group | 6 months
  Feasibility of recruiting as measured by the number of caregivers in the usual care who elect to receive the WLSCC protocol
Feasibility of training interventionist to deliver the WLSCC Intervention | 4 weeks
  Feasibility of interventionist training as measured by the number of hours required to prepare the interventionists
Fidelity to the intervention protocol | 6 months
  Fidelity rate as measured by the fidelity of intervention checklist
Feasibility of delivery of the WLSCC protocol by phone | 3 weeks
  Feasibility of delivering the WLSCC protocol by phone as measured by the rate of participation in phone calls
Feasibility of delivery duration of the WLSCC protocol by phone | 3 weeks
  Feasibility of delivering the WLSCC protocol by phone as measured by the duration of each phone call

SECONDARY OUTCOMES:
Cancer Caregiver Quality of Life [CQOLC] | 15 minutes
  35 items - 5-pt Likert scale; Sum of all item scores; higher scores mean better quality of life
Hospital Anxiety and Depression Scale (HADS) | 5 minutes
  7 on anxiety and 7 on depression; Sum of item scores on anxiety and depression; 11 and 21 "cases", 8 and 10 "borderline cases", and 0 and 7 as "non-cases"
Preparedness in Caregiving | 5 minutes
  8 items, 5-pt Likert scale (0 - 4); Sum of item scores divide by number of items; higher total score denotes higher preparedness
Multidimensional Scale of Perceived Social Support | 5 minutes
  7 pt Likert scale; Sum of item scores, then divide by number of items; higher score denotes higher perceived support
Functional Assessment of Cancer Therapy [FACT-G] | 15 minutes
  27 items, 5-point Likert scale; Sum of subscale scores; higher score, the better quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Cristina C Hendrix, DNS, GNP-BC, FAAN, Principal Investigator — Duke University School of Nursing
Locations (1):
- Duke Cancer Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No